CLINICAL TRIAL: NCT03059654
Title: Ultrasound-guided Percutaneous Dilatation Tracheostomy: Does it Have a Role in Obese Patients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohamed Emad El-Din Abdel-Ghaffar, Professor and chairman, department of Anesthesia and Intensive Care, Faculty of Medicine., Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: FOMSCU 2200
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Tracheostomy Techniques
Keywords: Percutaneous tracheostomy; surgical tracheostomy; airway ultrasound; intensive care
MeSH Terms: interventions — Tracheostomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound PCT (Active Comparator): Ultrasound guide Percutaneous tracheostomy
  Interventions: Procedure: tracheostomy
- Surgical tracheostomy (Active Comparator): Surgical tracheostomy
  Interventions: Procedure: tracheostomy

INTERVENTIONS:
Procedure: tracheostomy

SUMMARY:
To evaluate the usefulness of ultrasound-guided percutaneous dilatation tracheostomy PCT in obese patients.

DETAILED DESCRIPTION:
Aim of the work: to evaluate the usefulness of ultrasound-guided percutaneous dilatation tracheostomy PCT in obese patients.

Study objectives:

Primary: determine the duration of the procedure in both groups.

Secondary: determine the incidence of complications in both groups.

Setting of the study: This study will be conducted in the intensive care unit at Suez Canal University Hospital in Ismailia, Egypt.

Study design: prospective, randomized comparative clinical trial.

Sample size: At 95% level of confidence and 80% power of study, 30 patients per group will be sufficient to detect a difference of 15.1 ± 19.9 minutes between both groups using the following equation.

Where n= sample size

Z α/2 = 1.96 (The critical value that divides the central 95% of the Z distribution from the 5% in the tail)

Zβ = 0.84 (The critical value that separates the lower 20% of the Z distribution from the upper 80%)

σ = the estimate of the pooled standard deviation

µ1 = mean in the study group

µ2 = mean in the control group

(Bradley D., Karen I, et al, 2001)

Material and methods:

After obtaining the informed consent from patients' relatives the enrolled patients will be randomized into two study groups using table of random numbers:

1. Surgical tracheostomy (group S)
2. Ultrasound guided PCT (group U)

Past medical and surgical history will be taken from relatives of the patients. Examination of the site of skin incision for signs of infection or surgical or burn scars. Lab investigation will be done confirming that there is no coagulopathy (PT, INR, PTT and platelets)

Anesthesia will be achieved during the procedure with Propofol bolus of 1.5 - 2.5 mg / kg given intravenously. Analgesia will be provided by boluses of 1 µg / kg Fentanyl and relaxation will be achieved by 0.15 mg/kg Cis-atracurium intravenously if needed.

Patients will be ventilated with synchronized intermittent mandatory ventilation (SIMV) mode with FiO2 1.0 during the procedure.

The patients will be monitored continuously with heart rate, invasive blood pressure, 5-leads electrocardiogram, end-tidal capnogram and pulse oximetry (SpaO2).

The skin from the chin to the 3rd intercostals space will be sterilized with Povodine iodine 10% and the area around it will be covered with antiseptic drab.

Technique

In surgical tracheostomy group (group S):

The patient will be positioned in the supine position achieving hyperextension of the neck with roles behind the patient back.

An Ear-Nose-Throat surgeon will perform the surgical tracheostomy procedure after withdrawing the oral endotracheal tube to a level above the tracheostomy site.

The duration of the procedure will be estimated from the start of skin incision to the insertion of the tracheostomy tube into the trachea with confirmation by capnography and direct visualization of carina by bronchoscope though the tracheostomy tube.

In the ultrasound group (group U):

The patient position will be the same as done for surgical tracheostomy to achieve neck hyperextension. Two operators will perform the procedure, one will perform the ultrasound guided PCT and the other will visualize the procedure with fiber optic bronchoscope through the oral endotracheal.

An ultrasound examination of the anterior neck will be done identifying superficial veins, thyroid isthmus, cricoids, and tracheal cartilages to determine the site of needle puncture. After infiltrating the puncture site with Lidocaine 1% with Epinephrine 1:200,000 the catheter over needle will be advanced (in-plane) till it penetrates the anterior wall of the trachea using a 10-Heartz linear ultrasound probe (GE Healthcare, LOGIQ e ultrasound BT 12).

Next we will remove the needle leaving the catheter to introduce the J-guide wire after confirming the position of the needle visually by fiber optic bronchoscope and by aspiration of air through a saline syringe.

Then we will remove the ultrasound probe and the operator will pass the single beveled curved dilator (Blue Rhino) dilating the skin to the diameter required then the tracheostomy tube will be inserted into the trachea. Inflation of the tracheostomy will be done followed by connection of anesthetic breathing circuit confirming the proper position of the tracheostomy tube by capnography, chest expansion and lung sliding sign bilaterally.

For both groups the fiber optic bronchoscope will be also withdrawn from the oral endotracheal tube and reintroduced through the tracheostomy tube for detection of complications.

A chest X-ray will be obtained 3 hours later for confirmation of tracheostomy tube position and detection of early pneumothorax.

Data collection

The following data will be collected:

Gender, age (years), height (meters), weight (kilograms), body mass index (BMI) and the Sequential organ failure assessment (SOFA) will be recorded.

Heart rate, Blood pressure, SpaO2, End-tidal CO2 will be recorded every one minute. Anatomical landmark data in the form of trachea deviation, enlarged thyroid gland and apparent vessels at the puncture site will be recorded. Ultrasound data including tracheal deviation, level of the isthmus of thyroid gland, puncture site, subcutaneous vessels, the tracheal diameter (centimeters) and skin-to-anterior tracheal thickness (centimeters) will be recorded.

In (group S) the duration of the procedure will be timed from the start of land mark identification to the insertion of the tracheostomy tube and in (group U) the duration of the procedure will be timed from the start of ultrasound examination of the neck to the insertion of the tracheostomy tube (measured in minutes).

Early complication such as esophageal injury, posterior tracheal wall injury, massive bleeding, tracheostomy malpositioning, hypoxemia (pulse oximetry < 90%), hypotension (systolic blood pressure < 90 mmHg, tracheal cuff puncture and tracheal ring fractures will be recorded. Also late complications such as tracheal subglottic stenosis, stomal infection, pneumothorax and subcutaneous emphysema will be recorded.

Ethical consideration

* The ultrasound technology has been used in anesthesia and intensive care successfully and it is non-invasive facilitating most procedures done in both fields especially in obese patients.
* A written informed consent will be obtained from the patients or patients' relatives before being involved in the study.
* The steps of the study; the aims, the benefits and disadvantages, all will be discussed with the patients or patients' relatives.
* The patient has the right to refuse participation.
* Any abnormal results will be managed according to traditional methods.
* Confidentiality of all data and test results of all the study population are preserved.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill patients aged over 18 years old needing tracheostomy.
2. Both genders.
3. Obese patients with neck circumference ≥ 40 cm.

Exclusion Criteria:

1. Patients with coagulopathy (partial thromboplastin time > 50 seconds and international normalization ratio > 1.5 or platelets count < 80000 / mm3).
2. History of difficult laryngoscopy (Cormack-Lehane Grade 2b view) documented on intubation.
3. Requirement of high Positive End Expiratory Pressure (PEEP > 10 cmH2O) or high fraction inspired oxygen (FiO2 > 0.8).
4. Infection at the site of tracheostomy.
5. Previous neck surgery or radiotherapy.
6. Hypersensitivity to local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Duration of the procedure in both groups in minutes | average forty five minutes.
  From start of procedure till skin closure

SECONDARY OUTCOMES:
incidence of complications in both groups | four weeks
  From start of procedure till hospital discharge or death.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Suez Canal University Hospital, Ismailia, Ismailia Governorate
  - Suez Canal University hospital, Ismailia, Ismailia Governorate